CLINICAL TRIAL: NCT00882544
Title: Prospective Pediatric Pyeloplasty Robotic Surgical Database
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-112
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hydronephrosis
Keywords: hydronephrosis; robotic pyeloplasty; pediatric pyeloplasty
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosed Pediatric Hydronephrosis: Children diagnosed with hydronephrosis who are to receive robotic pyeloplasty surgery

SUMMARY:
Performance and outcomes measure are, at this time, relatively unknown for robotic pyeloplasty procedures. The purpose of this study is to provide a clearer understanding of the urology department's robotic pyeloplasty quality and outcomes measures. This will be accomplished by prospectively collecting data for these procedures would ensure that measures are consistently collected in accordance with a defined protocol, allowing for more valuable quality and clinical research analysis.

Hypothesis will be defined before data analysis is performed. Amendments specifying future hypothesis will be submitted the IRB at the appropriate time.

DETAILED DESCRIPTION:
Minimally invasive surgery is becoming a widely accepted method of surgery for many urological conditions. This includes both laparoscopy and robotic assisted laparoscopic surgery. In adult urology, there is discussion of laparoscopic pyeloplasty replacing open surgery as the gold standard in the treatment of ureteropelvic junction obstruction. Although at a slower rate, minimally invasive surgery is also becoming a standard method of treatment in the pediatric setting. Some urological surgeons are predicting that laparoscopy will become the standard of treatment in the straightforward pediatric nephrectomy. Benefits of laparoscopic surgery include improved cosmesis, reduced postoperative pain issues, and reduced length of stay. However, laparoscopic use for more delicate or complicated procedures has been limited due to 2-dimensional imaging, rigid non-articulating instruments, and the time and expense required for surgeons to master these techniques.

The advent of robotic surgery minimizes or eliminates many of these issues. Hand and wrist movements with the robot more closely mimic the actual hand and wrist movements in open surgery. Three-dimensional imaging provides the surgeon with necessary depth perception, articulating instruments with six degrees of freedom allow the surgeon to tie knots and suture more easily, and the learning curve has been reduced. Robotic surgery has the added benefit over laparoscopy with the introduction of tremor-filtering instruments and movement scaling. As of 2006, there were about 400 robots worldwide, and most were used primarily for urological surgery.

Currently, the most common procedure in pediatric robotic surgery is pyeloplasty, followed by fundoplication, and patent ductus arteriosus ligation. However, robotic surgery can be used in more difficult reconstructive surgeries, such as appendicovesicostomy and bladder augmentation in the pediatric population. The major impediment to widespread applications of minimally invasive surgery in pediatric procedures has been laparoscopic suturing. With increased accuracy, the advent of smaller instruments, and three-dimensional imaging, robotics is now a premier surgical advancement, and has allowed minimally invasive surgery to become a viable treatment method to a wider range of procedures and surgeons.

The first report of pediatric robotic surgery was published in 2002 and described successful surgeries of fundoplication, cholecystectomy, and salpingoophorectomy using the da Vinci robotic system. Two recent literature reviews of pediatric robotic surgery report that the majority of studies published in this area are either case report or case series.6 , One of the systematic reports was published in Spanish, so only the translated abstract was available to this department. The second systematic review reported that as of October 2007, there were 31 studies published describing 566 patients. Only four studies were case control, comparing robotic surgery with either laparoscopic or open procedures. Two of these case control reports described robotic assisted pyeloplasty in children compared to open surgery. As can be seen from these meta-analysis, published studies on robotic surgery is in its infancy and additional studies are necessary.

The purpose of this research is to provide a clearer understanding of the urology department's robotic pyeloplasty quality and outcomes measures. This will be accomplished by developing a database for research.

Specific Aim 1: To consistently collect performance and outcomes data for robotic pyeloplasty procedures in order to increase internal understanding of these procedures.

Specific Aim2: To consistently collect performance and outcomes data for robotic pyeloplasty procedures in order to perform more valuable clinical analysis for publication.

Hypothesis will be defined before data analysis is performed. Amendments specifying future hypothesis will be submitted the IRB at the appropriate time.

ELIGIBILITY:
Inclusion Criteria:

* Subject received a robotic pyeloplasty procedure at Connecticut Children's Medical Center
* Subject signs informed consent and HIPAA Authorization

Exclusion Criteria:

* Subject did not receive a robotic pyeloplasty procedure at Connecticut Children's Medical Center
* Subject does not sign informed consent and/or HIPAA Authorization

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 0-18 years of age who receive a robotic pyeloplasty procedure at Connecticut Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Resolution of Hydronephrosis | 3 to 6 months after surgical intervention

SECONDARY OUTCOMES:
Symptom Resolution at follow-up | 3 to 6 months after surgical intervention
Drainage at Follow-up by MAG3 | 3 to 6 months after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katherine W Herbst, M.Sc, Study Director — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon DA, El-Shazly MA, Chang CM, Gianduzzo TR, Eden CG. Laparoscopic pyeloplasty: evolution of a new gold standard. Urology. 2006 May;67(5):932-6. doi: 10.1016/j.urology.2005.11.024. Epub 2006 Apr 25. PMID 16635516
- [Background] Smaldone MC, Sweeney DD, Ost MC, Docimo SG. Laparoscopy in paediatric urology: present status. BJU Int. 2007 Jul;100(1):143-50. doi: 10.1111/j.1464-410X.2007.06854.x. Epub 2007 Apr 5. PMID 17419701
- [Background] Chacko JK, Koyle MA, Mingin GC, Furness PD 3rd. Minimally invasive open renal surgery. J Urol. 2007 Oct;178(4 Pt 2):1575-7; discussion 1577-8. doi: 10.1016/j.juro.2007.05.099. Epub 2007 Aug 16. PMID 17707048
- [Background] Meehan JJ, Meehan TD, Sandler A. Robotic fundoplication in children: resident teaching and a single institutional review of our first 50 patients. J Pediatr Surg. 2007 Dec;42(12):2022-5. doi: 10.1016/j.jpedsurg.2007.08.022. PMID 18082700
- [Background] Menon M, Hemal AK. Robotic urologic surgery: is this the way of the future? World J Urol. 2006 Jun;24(2):119. doi: 10.1007/s00345-006-0081-3. No abstract available. PMID 16622692
- [Background] Passerotti C, Peters CA. Robotic-assisted laparoscopy applied to reconstructive surgeries in children. World J Urol. 2006 Jun;24(2):193-7. doi: 10.1007/s00345-006-0084-0. No abstract available. PMID 16758249
- [Background] Lee RS, Borer JG. Robotic surgery for ureteropelvic junction obstruction. Curr Opin Urol. 2006 Jul;16(4):291-4. doi: 10.1097/01.mou.0000232052.74342.a0. PMID 16770130
- [Background] Gutt CN, Markus B, Kim ZG, Meininger D, Brinkmann L, Heller K. Early experiences of robotic surgery in children. Surg Endosc. 2002 Jul;16(7):1083-6. doi: 10.1007/s00464-001-9151-1. Epub 2002 Apr 9. PMID 12165827
- [Background] Estrada CR, Passerotti CC. [Robotic surgery in pediatric urology]. Arch Esp Urol. 2007 May;60(4):471-9. doi: 10.4321/s0004-06142007000400017. Spanish. PMID 17626539